CLINICAL TRIAL: NCT01185132
Title: A Phase III Randomized Study Comparing Intensity Modulated Planning Versus 3-Dimensional Planning for Accelerated Partial Breast Radiotherapy
Brief Title: Intensity Modulated Radiotherapy (IMRT) vs. 3D-conformal Accelerated Partial Breast Irradiation (APBI) for Early Stage Breast Cancer After Lumpectomy
Acronym: 2009-APBI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rocky Mountain Cancer Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-APBI; WIRB #20091193 (Other: Western IRB)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: breast-conservation; adjuvant radiotherapy; breast cancer; early-stage breast cancer; DCIS; lumpectomy; accelerated partial breast irradiation; APBI; three dimensional conformal external radiotherapy; intensity modulated radiotherapy; 3D CRT; IMRT
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMRT (Experimental): Intensity modulated radiotherapy, 38.5 Gy, 10 fractions over 5 days
  Interventions: Radiation: accelerated partial breast irradiation - IMRT planning
- 3D-CRT (Active Comparator): Three dimensional conformal external radiotherapy, 38.5 Gy, 10 fractions over 5 days
  Interventions: Radiation: accelerated partial breast irradiation - 3D-conformal planning

INTERVENTIONS:
Radiation: accelerated partial breast irradiation - 3D-conformal planning — 38.5 Gy, 10 fractions over 5 days
  Other Names: APBI; EBRT
  Arms: 3D-CRT
Radiation: accelerated partial breast irradiation - IMRT planning — 38.5 Gy, 10 fractions over 5 days
  Other Names: APBI; EBRT
  Arms: IMRT

SUMMARY:
In the setting of radiotherapy as part of breast-conservation therapy for patients with early stage breast cancer, the novel planning and delivery method of intensity modulated radiotherapy is an effective and safe alternative to the commonly-used standard 3D-conformal external beam radiotherapy, spares more normal breast and lung tissue, and may lead to improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed disease (AJC Classification): Tis, T1, T2 (≤ 3.0 cm), N0, M0.
* Microscopic multifocal disease is only allowed when the entire span of identified disease measures 3.0 cm or less.
* Negative surgical margins ( ≥ 0.2 cm) after final surgery.
* Subjects with infiltrating lobular histologies or high nuclear grade DCIS will be required to have breast MRI scanning as part of the initial staging to verify localized disease.
* Subjects with DCIS will be included in the study only if they had an MRI prior to lumpectomy.
* Findings on MRI scanning revealing relevant suspicion of disease outside of planned lumpectomy volume should be further evaluated by ultrasound and, if necessary biopsy, to exclude multicentric/multifocal disease.
* Subjects with malignant calcifications on mammography will be required to have repeat mammography after surgery to ensure removal of all malignant calcifications.
* Willing to complete additional screening requirements and meet eligibility criteria as defined in protocol Sec. 4.4.
* Successful placement of fiducial markers for IGRT requiring nonmigrating fiducials.
* PTV to ipsilateral breast ratio (IBR) ≤ 25 %.
* Radiotherapy anticipated to begin within 10 weeks of lumpectomy or re-excision of margins.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Have collagen-vascular disease.
* Inadequate surgical margins ( < 0.2 cm) after final surgery.
* Subjects with persistent malignant/suspicious micro-calcifications.
* Gross multifocal disease and microscopic disease greater than 3.0 cm.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2009-07; Primary Completion 2018-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of breast pain after Accelerated Partial Breast Radiotherapy (APBI) | 5 years
  Assessment by both treating investigators and by subjective patient outcomes questionnaires filled out at each follow-up visit
Prevalence of chest wall pain after Accelerated Partial Breast Radiotherapy (APBI) | 2-5 years
  Assessment by both treating investigators and by subjective patient outcomes questionnaires filled out at each follow-up visit

SECONDARY OUTCOMES:
Dosimetric comparison | 5-10 days
  Comparison of treatment plans and actual doses received between comparable patients treated with 3D-CRT and IMRT with regard to treatment target and normal tissue
Acute skin reactions | 6 months
  Radiation-induced dermatitis
Cosmetic outcomes after APBI | 2-5 years
  Assesed by both treating investigators and subjective patient questionnaires filled out at each follow-up visit
Ipsilateral breast event | 5-15 years
  Track occurrence and patterns of local treatment failures or new primaries within the treated breast (efficacy outcome measure)
Cause specific survival | 5-15 years
  Track survival status and the specific cause(s) of death if applicable for study participants (efficacy outcome measure)
Disease free survival | 5-15 years
  Track breast-cancer free survival status of study participants (efficacy outcome measure)
Overall survival | 5-15 years
  Track the overall survival status of all study participants (efficacy outcome measure)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Leonard, MD, Principal Investigator — Rocky Mountain Cancer Centers
Locations (5):
- United States (5):
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado

REFERENCES:
- [Derived] Leonard CE, Wang Y, Asmar L, Lei RY, Howell KT, Henkenberns PL, Johnson TK, Hobart TL, Tole SP, Kercher JM, Widner JL, Barke L, Kaske T, Carter DL. A prospective Phase III trial evaluating patient self-reported pain and cosmesis in accelerated partial breast irradiation utilizing 3-D versus intensity-modulated radiotherapy. Cancer Med. 2021 Oct;10(20):7089-7100. doi: 10.1002/cam4.4242. Epub 2021 Sep 1. PMID 34469056